CLINICAL TRIAL: NCT01984801
Title: A Single-Blind Study to Evaluate the Irritation Potential of Repeat Topical Applications of GSK1940029 Gel on the Intact Skin of Healthy Human Subjects and Acne Patients
Brief Title: Study to Investigate the Irritation Potential of GSK1940029 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 117225
Record Dates: First submitted 2013-09-05; First posted 2013-11-15 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
Keywords: SCD1; Gel; Topical Administration; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — long-chain-aldehyde dehydrogenase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Each of the following 6 treatments will be randomized to one of 6 designated locations on either upper arm or other locations, such as the lower or upper back, within each healthy subject: (A) 200 mg of 0.3% GSK1940029 gel, (B) 200 mg of 1% GSK1940029 gel, (C) 200 mg of 0.3%/1% vehicle gel only, (D) 200 µL of sterile distilled water, (E) Patch only, and (F) 200 µL of 0.5% SLS in sterile distilled water, Each treatment will be applied using individual patches, daily for 2 days
  Interventions: Drug: 0.3% GSK1940029 gel; Drug: 1% GSK1940029 gel; Drug: 0.3%/1% vehicle gel only; Other: Sterile distilled water; Other: 0.5% SLS in sterile distilled water; Other: Patch only
- Part 2 (Experimental): Each of the following 6 treatments will be randomized to one of 6 designated locations on either upper arm or other locations, such as the lower or upper back, within each healthy subject: (A) 200 mg of 0.3% GSK1940029 gel, (B) 200 mg of 1% GSK1940029 gel, (C) 200 mg of 0.3%/1% vehicle gel only, (D) 200 µL of sterile distilled water, (E) Patch only, and (F) 200 µL of 0.1% SLS in sterile distilled water. Each treatment will be applied using individual patches, daily for 21 days
  Interventions: Drug: 0.3% GSK1940029 gel; Drug: 1% GSK1940029 gel; Drug: 0.3%/1% vehicle gel only; Other: Sterile distilled water; Other: 0.1% SLS in sterile distilled water; Other: Patch only
- Part 3 (Experimental): Each acne patient will apply a thin coat of one or two concentration of GSK1940029 gel or vehicle to acne affected facial/neck skin by hand, once daily for 28 days
  Interventions: Drug: 0.3% GSK1940029 gel; Drug: 1% GSK1940029 gel; Drug: 0.3%/1% vehicle gel only

INTERVENTIONS:
Drug: 0.3% GSK1940029 gel — 200 mg of the gel will be applied to individual patches by using a spatula
Drug: 1% GSK1940029 gel — 200 mg of the gel will be applied to individual patches by using a spatula
Drug: 0.3%/1% vehicle gel only — 200 mg of the gel will be applied to individual patches by using a spatula
Other: Sterile distilled water — 200 µL of the solution will be applied to individual patches by using a pipette or syringe
  Arms: Part 1; Part 2
Other: 0.5% SLS in sterile distilled water — 200 µL of the solution will be applied to individual patches by using a pipette or syringe
  Arms: Part 1
Other: 0.1% SLS in sterile distilled water — 200 µL of the solution will be applied to individual patches by using a pipette or syringe
  Arms: Part 2
Other: Patch only — Only patch will be applied
  Arms: Part 1; Part 2

SUMMARY:
The proposed indication for GSK1940029 is topical treatment of acne, the early clinical plan will evaluate the irritation potential of GSK1940029 (Study SCD117225 - 3 Part study); and safety, tolerability and pharmacokinetics of GSK1940029 (Study SCD117226 - 2 Part study), after topical administration on healthy subjects and acne patients. Study SCD117225 will be a randomized, single-blind, three part study, to evaluate the primary irritation potential (Part 1), cumulative irritation potential (Part 2) of two concentrations of GSK1940029 gel applied to the intact skin of healthy subjects, and the facial irritation potential of one or two concentrations of GSK1940029 applied to the face of acne patients (Part3). In Part 1 and Part 2 the following 6 treatments will be applied using individual patches: (A) 200 milligrams (mg) of 0.3% GSK1940029 gel, (B) 200 mg of 1% GSK1940029 gel, (C) 200 mg of 0.3%/1% vehicle gel only (vehicle control), (D) 200 microliters (µL) of sterile distilled water (negative irritant control), (E) 200 µL of - 0.5% sodium lauryl sulfate (SLS) in sterile distilled water for Part 1/0.1% SLS in sterile distilled water for Part 2 (positive irritant control), and (F) Patch only (patch control). Each treatment will be randomized to one of six designated locations on either upper arm or other locations, such as the lower or upper back, within each subject. The same treatment will be reapplied to the same location on subsequent days. Each treatment will be applied daily for 2 days in Part 1, and daily for 21 days in Part 2. In Part 3, each patient will apply a thin coat of one or two concentration of GSK1940029 gel or vehicle to acne affected facial/neck skin by hand, once daily for 28 days. Parts within Study SCD117225 and Study SCD117226 will have interdependencies. No significant primary irritation signal in Study SCD117225 Part 1 would allow initiation of Study SCD117226 Part 1 (single dose application). Once safety, tolerability and exposure information are determined in Study SCD117226 Part 1, Part 2 of Study SCD117225 may be initiated along with Part 2 (14-day repeat dose application). No significant cumulative irritation signal (study SCD117225 Part 2) in combination with adequate 14-day safety (study SCD117226 Part 2) would allow initiation of Part 3 of Study SCD117225.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring for Parts 1 and 2 only.
* Moderate/Moderate to Severe acne patients, otherwise healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring for Part 3 only.
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international units (MIU)/millilitres (mL) and estradiol <40 picograms (pg)/mL (<147 picomoles [pmol]/liter [L]) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will not be allowed.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until after study follow-up visit.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged assessments, QT duration corrected for heart rate (QTc) <450 msec; or QTc <480 msec in subjects with bundle branch block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome for all study Parts and asymptomatic gallstones for Parts 1 and 2 only). Subjects with a history of gall stones, asymptomatic gallstones or cholecystectomy will be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 standard drinks. One standard drink is equivalent to 10 grams (g) of alcohol: 285 mL of beer, 100 mL of wine or 30 mL of 40% alcohol by volume distilled spirits.
* History of or current meibomian gland dysfunction or dry eye disease
* History or presence of significant skin disorder (such as but not limited to severe (extensive) atopic dermatitis, severe eczema, psoriasis or skin cancer) that would in any way confound interpretation of the study results, or subjects who present with damaged skin including sunburn, moles, uneven skin tones, scar tissue, tattoos, body piercings, sunburn, branding or other disfiguration on or near the intended site of application which could interfere with the grading. Acne is allowed for Part 3.
* History of cutaneous photodisorder, such as photoallergic reaction or polymorphic light eruption. History of cold urticaria and reactions to extreme temperatures.
* History of allergy to soaps, lotions, cosmetics, tape/adhesives, petrolatum or latex or topical drugs of same class as the study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of severe, chronic asthma or significant allergies (including food, drug or cutaneous allergies). Subjects with the presence or a history of atopy (seasonal allergies, allergic rhinitis) or mild (limited) eczema will be allowed to participate in the study, although applications at sites with active eczema will not be allowed.
* Use of topical medications such as but not limited to retinoids, steroids, and transdermal hormone replacement therapies on or near the intended site of application within 8 weeks prior to dosing through treatment follow up, for Parts 1 and 2 only or within 2 weeks period to dosing for Part 3. Use of other topical preparations such as those containing vitamins, supplements or herbal within 2 weeks prior to dosing through treatment follow up.
* Unable to refrain from the use of topical medications from the initial dose of study medication through follow-up.
* Foreseeable intensive Ultraviolet (UV) exposure during the study (solar or artificial) as follows: subjects must not be exposed to direct sunlight for sun tanning or exposed to skin tanning devices (e.g. sunbed) for the duration of the study.
* Participation in any patch test for cumulative irritation or sensitization within 4 weeks preceding the first dose of study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2015-04-10 (Actual)

PRIMARY OUTCOMES:
Primary cutaneous irritation scores | Days 2, 3 4 and 5 of Part 1
  The patch/test sites will be evaluated for irritation potential and will be graded using a grading scale based on scales developed by Hill Top Research, Inc and cited by the United States (US) Food and Drug Administration (FDA) in the Draft Guidance for Industry: Skin Irritation and Sensitization Testing of Generic Transdermal Drug Products, December 1999
Cumulative cutaneous irritation scores | Day 2 to Day 22 of Part 2
  Visual evaluations of the patch/test sites will be performed for irritation potential approximately 24 hours after each patch application, and will be graded using a grading scale based on scales developed by Hill Top Research, Inc and cited by the US FDA in the Draft Guidance for Industry: Skin Irritation and Sensitization Testing of Generic Transdermal Drug Products, December 1999
Facial irritation scores | Days 1, 7, 14, 21, 28, 29 and at FU (Days 35-42) of Part 3
  The Facial Irritation Scoring System will be based on the Draize Scoring System with an additional Sensation of Burning/Stinging category
Lanman-Maibach irritation classifications | Day 2 to Day 22 of Part 2
  The derived cumulative irritation scores will be interpreted using the Lanman-Maibach classification system
Tolerability of GSK1940029 as assessed by Clinical monitoring/observation | Up to Day 17 of Part 1, Up to Day 36 of Part 2, and Up to Day 42 of Part 3
Tolerability of GSK1940029 as assessed by adverse events (AEs) | Up to Day 17 of Part 1, Up to Day 36 of Part 2, and Up to Day 42 of Part 3

SECONDARY OUTCOMES:
Safety and tolerability of GSK1940029 as assessed by clinical laboratory tests | Screening, Days 1, 4, and FU (Days 10 to 17) of Part 1. Screening, Days 1, 8, 22, and FU (Days 29 to 36) of Part 2. Screening, Days 1, 7, 14, 21, 29, and FU (Days 35 to 42) of Part 3.
  Clinical laboratory tests will include hematology, chemistry and urinalysis parameters
Safety and tolerability of GSK1940029 as assessed by vital signs measurements | Screening, Days 1, 2, and FU (Days 10 to 17) of Part 1. Screening, Days 1, 2 and FU (Days 29 to 36) of Part 2. Screening, Days 1, 2 and FU (Days 35 to 42) of Part 3
  Vital signs measurements will include systolic and diastolic blood pressure and heart rate
Safety and tolerability of GSK1940029 as assessed by clinical monitoring/observation | Up to Day 17 of Part 1, Up to Day 36 of Part 2, and Up to Day 42 of Part 3
Ocular tolerability of topical applications of GSK1940029 | Screening, Days 1, 5, and FU (Days 10 to 17) of Part 1. Screening, Days 1, 22, and FU (Days 29 to 36) of Part 2. Screening, Days 1, 7, 14, 21, 29, and FU (Days 35 to 42) of Part 3.
  Eye examination will be performed. Ocular evaluations will include slit lamp examination with fluorscein, tear film breakup time, visual acuity and ocular surface disease index
Plasma GSK1940029 pharmacokinetics (PK) | Part 3 Only - Days 1 and 28: pre-dose, 2, 4, and 8 hours post-dose; Day 2: pre-dose; and Day 29: 24 hour post-Day 28 dose
  Blood samples for PK analysis of GSK1940029 will be collected. PK parameters will include Area under the concentration-time curve: from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments [AUC(0-t)] and from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)]; maximum observed concentration (Cmax); time of occurrence of cmax (tmax); and terminal phase half-life (t1/2) as data permit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- See also: Results for study 117225 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117225?search=study&study_ids=117225#rs